CLINICAL TRIAL: NCT00005153
Title: Etiologic Risk Factors of Cardiovascular Malformations
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1025; R37HL025629 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2001-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Defect, Congenital Heart
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Defects, Congenital

SUMMARY:
To identify genetic and environmental risk factors for congenital cardiac disease.

DETAILED DESCRIPTION:
BACKGROUND:

Congenital heart disease represents a major segment of clinically significant birth defects and is associated with high mortality and morbidity in infancy, a childhood marred with physical limitations and repeated invasive procedures, and an adulthood with increased risk of medical and social problems. Previous research has been principally directed to clinical methods of diagnosis and treatment, but the need for prediction and prenatal counseling requires further knowledge of environmental and familial risk factors. Congenital heart disease is not one of the malformations monitored by the International Clearing House of Birth Defects Surveillance System. Surveillance which does include congenital heart disease may lack diagnostic accuracy among the various reporting sources. Accurate clinical studies lack comparative control information. As a result, the true epidemiologic features of cardiac defects remain obscure.

DESIGN NARRATIVE:

The design of the Baltimore-Washington Infant Study was that of a case-control study. All infants under one year of age with confirmed diagnoses of congenital heart disease were eligible for inclusion if they were residents of the study area which encompassed 53 area hospitals in Maryland, the District of Columbia and five counties in Virginia. Case enrollment was done through five pediatric cardiology centers and through a periodic search of the obstetrics and neonatal and pathology logs of the participating hospitals. Control selection was by random numbers and all resident births were eligible as controls except for those with congenital heart disease. Mothers of cases and controls were interviewed at home for demographic information, and information on maternal health, maternal medication, reproductive history, lifestyle, environmental exposures in the home, occupation, and agents transmitted to the mother by the father. Data were collected on the characteristics, drug use, habits, and occupations of the fathers. Vital records and birth certificates were abstracted for all cases and controls. Death certificates were also abstracted. Variables including drugs, lifestyle and home exposures, and occupation, were screened to identify which single factors were most importantly related to congenital heart disease.

Cases in which congenital heart disease was part of a genetic complex were evaluated separately for environmental exposures. Genetic data analysis focused on first degree relatives but extended family data were noted wherever available. The genetic data analyses included: estimation of recurrence risks in siblings for congenital heart disease with the same cardiac defect; any cardiac defect in the sibling; non cardiac birth defect and pregnancy loss in the family. Parental phenotype was investigated for the presence of birth defects and known genetic disorders. Twin births were assessed for concordance in zygosity. Hypotheses of genetic and environmental teratogenic and coteratogenic interactions were tested. Pathogenic mechanisms were further defined through anatomic and echocardiographic observations. The family inquiry was expanded to include cousins. Nutrition information was added on maternal vitamin A supplementation, protein, calories, and other nutrients.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1980-12; Study Completion 1998-11 (Actual)

REFERENCES:
- [Background] Scanlon KS, Ferencz C, Loffredo CA, Wilson PD, Correa-Villasenor A, Khoury MJ, Willett WC. Preconceptional folate intake and malformations of the cardiac outflow tract. Baltimore-Washington Infant Study Group. Epidemiology. 1998 Jan;9(1):95-8. PMID 9430276
- [Background] Lurie IW, Ferencz C. VACTERL-hydrocephaly, DK-phocomelia, and cerebro-cardio-radio-reno-rectal community. Am J Med Genet. 1997 May 16;70(2):144-9. doi: 10.1002/(sici)1096-8628(19970516)70:23.0.co;2-y. PMID 9128933
- [Background] Lurie IW, Kappetein AP, Loffredo CA, Ferencz C. Non-cardiac malformations in individuals with outflow tract defects of the heart: the Baltimore-Washington Infant Study (1981-1989). Am J Med Genet. 1995 Oct 23;59(1):76-84. doi: 10.1002/ajmg.1320590116. PMID 8849016
- [Background] Teratogenicity of progestational agents. Teratology. 1984 Feb;29(1):131-46. doi: 10.1002/tera.1420290115. No abstract available. PMID 6701803
- [Background] Ferencz C, Rubin JD, McCarter RJ, Wilson PD, Brenner JI, Neill CA, Perry LW, Hepner SI, Downing JW: Association of Blood Disorders and Congenital Heart Disease (Letter). Teratology, 29(2):313, 1984
- [Background] Ferencz C, Rubin JD, McCarter RJ, Wilson PD, Boughman JA, Brenner JI, Neill CA, Perry LW, Hepner SI, Downing JW. Hematologic disorders and congenital cardiovascular malformations: converging lines of research. J Med. 1984;15(5-6):337-54. PMID 6399520
- [Background] Ferencz C, Rubin JD, McCarter RJ, Brenner JI, Neill CA, Perry LW, Hepner SI, Downing JW. Congenital heart disease: prevalence at livebirth. The Baltimore-Washington Infant Study. Am J Epidemiol. 1985 Jan;121(1):31-6. doi: 10.1093/oxfordjournals.aje.a113979. PMID 3964990
- [Background] Ferencz C, Rubin JD, McCarter RJ, Brenner JI, Neill CA, Perry LW, Hepner SI, Downing JW. Maternal mitral valve prolapse and congenital heart disease in the offspring. Am Heart J. 1985 Oct;110(4):899-900. doi: 10.1016/0002-8703(85)90483-1. No abstract available. PMID 4050668
- [Background] Kaden GG, McCarter RJ, Johnson SF, Ferencz C. Physician-patient communication. Understanding congenital heart disease. Am J Dis Child. 1985 Oct;139(10):995-9. doi: 10.1001/archpedi.1985.02140120041025. PMID 4036904
- [Background] Rubin JD, Ferencz C, McCarter RJ, Wilson PD, Boughman JA, Brenner JI, Neill CA, Perry LW, Hepner SI, Downing JW. Congenital cardiovascular malformations in the Baltimore-Washington area. Md Med J. 1985 Nov;34(11):1079-83. No abstract available. PMID 3853721
- [Background] Rubin JD, Ferencz C. Subsequent pregnancy in mothers of infants with congenital heart disease. Pediatrics. 1985 Sep;76(3):371-4. PMID 4034297
- [Background] Ferencz C. The etiology of congenital cardiovascular malformations: observations on genetic risks with implications for further birth defects research. J Med. 1985;16(5-6):497-508. PMID 2937867
- [Background] Ferencz C. Offspring of fathers with cardiovascular malformations. Am Heart J. 1986 Jun;111(6):1212-3. doi: 10.1016/0002-8703(86)90034-7. No abstract available. PMID 3716999
- [Background] Boughman JA, Berg KA, Astemborski JA, Clark EB, McCarter RJ, Rubin JD, Ferencz C. Familial risks of congenital heart defect assessed in a population-based epidemiologic study. Am J Med Genet. 1987 Apr;26(4):839-49. doi: 10.1002/ajmg.1320260411. PMID 3591826
- [Background] Johnson SF, McCarter RJ, Ferencz C. Changes in alcohol, cigarette, and recreational drug use during pregnancy: implications for intervention. Am J Epidemiol. 1987 Oct;126(4):695-702. doi: 10.1093/oxfordjournals.aje.a114709. PMID 3498364
- [Background] Ferencz C, Rubin JD, McCarter RJ, Boughman JA, Wilson PD, Brenner JI, Neill CA, Perry LW, Hepner SI, Downing JW. Cardiac and noncardiac malformations: observations in a population-based study. Teratology. 1987 Jun;35(3):367-78. doi: 10.1002/tera.1420350311. PMID 3629517
- [Background] Boughman JA, Astemborski JA, Berg KA, Clark EB, Ferencz C. Variation in expression of congenital cardiovascular malformations within and among families. Basic Life Sci. 1988;43:93-103. doi: 10.1007/978-1-4684-5460-4_10. No abstract available. PMID 3365227
- [Background] Wilson PD, Ferencz C, Dischinger PC, Brenner JI, Zeger SL. Twenty-four-hour ambulatory blood pressure in normotensive adolescent children of hypertensive and normotensive parents. Am J Epidemiol. 1988 May;127(5):946-54. doi: 10.1093/oxfordjournals.aje.a114898. PMID 3358415
- [Background] Maestri NE, Beaty TH, Liang KY, Boughman JA, Ferencz C. Assessing familial aggregation of congenital cardiovascular malformations in case-control studies. Genet Epidemiol. 1988;5(5):343-54. doi: 10.1002/gepi.1370050505. PMID 3215508
- [Background] Ferencz C, Neill CA, Boughman JA, Rubin JD, Brenner JI, Perry LW. Congenital cardiovascular malformations associated with chromosome abnormalities: an epidemiologic study. J Pediatr. 1989 Jan;114(1):79-86. doi: 10.1016/s0022-3476(89)80605-5. PMID 2521249
- [Background] Ferencz C. Origin of congenital heart disease: reflections on Maude Abbott's work. Can J Cardiol. 1989 Jan-Feb;5(1):4-9. PMID 2645982
- [Background] Ferencz C, Boughman JA, Neill CA, Brenner JI, Perry LW. Congenital cardiovascular malformations: questions on inheritance. Baltimore-Washington Infant Study Group. J Am Coll Cardiol. 1989 Sep;14(3):756-63. doi: 10.1016/0735-1097(89)90122-8. PMID 2768723
- [Background] Martin GR, Perry LW, Ferencz C. Increased prevalence of ventricular septal defect: epidemic or improved diagnosis. Pediatrics. 1989 Feb;83(2):200-3. PMID 2783625
- [Background] Berg KA, Astemborski JA, Boughman JA, Ferencz C. Congenital cardiovascular malformations in twins and triplets from a population-based study. Am J Dis Child. 1989 Dec;143(12):1461-3. doi: 10.1001/archpedi.1989.02150240083023. PMID 2589279
- [Background] Ferencz C, Rubin JD, McCarter RJ, Clark EB. Maternal diabetes and cardiovascular malformations: predominance of double outlet right ventricle and truncus arteriosus. Teratology. 1990 Mar;41(3):319-26. doi: 10.1002/tera.1420410309. PMID 2326756
- [Background] Ferencz C. On the birth prevalence of congenital heart disease. J Am Coll Cardiol. 1990 Dec;16(7):1701-2. doi: 10.1016/0735-1097(90)90322-g. No abstract available. PMID 2254556
- [Background] Carmi R, Boughman JA. Pentalogy of Cantrell and associated midline anomalies: a possible ventral midline developmental field. Am J Med Genet. 1992 Jan 1;42(1):90-5. doi: 10.1002/ajmg.1320420118. PMID 1308371
- [Background] Carmi R, Boughman JA, Ferencz C. Endocardial cushion defect: further studies of "isolated" versus "syndromic" occurrence. Am J Med Genet. 1992 Jun 1;43(3):569-75. doi: 10.1002/ajmg.1320430313. PMID 1534968
- [Background] Ferencz C, Neill CA. Cardiomyopathy in infancy: observations in an epidemiologic study. Pediatr Cardiol. 1992 Apr;13(2):65-71. doi: 10.1007/BF00798206. PMID 1614921
- [Background] Correa-Villasenor A, Ferencz C, Boughman JA, Neill CA. Total anomalous pulmonary venous return: familial and environmental factors. The Baltimore-Washington Infant Study Group. Teratology. 1991 Oct;44(4):415-28. doi: 10.1002/tera.1420440408. PMID 1962287
- [Background] Correa-Villasenor A, McCarter R, Downing J, Ferencz C. White-black differences in cardiovascular malformations in infancy and socioeconomic factors. The Baltimore-Washington Infant Study Group. Am J Epidemiol. 1991 Aug 15;134(4):393-402. doi: 10.1093/oxfordjournals.aje.a116101. PMID 1877600
- [Background] Rosenthal GL, Wilson PD, Permutt T, Boughman JA, Ferencz C. Birth weight and cardiovascular malformations: a population-based study. The Baltimore-Washington Infant Study. Am J Epidemiol. 1991 Jun 15;133(12):1273-81. doi: 10.1093/oxfordjournals.aje.a115839. PMID 2063835
- [Background] Lurie IW, Magee CA, Sun CC, Ferencz C. 'Microgastria--limb reduction' complex with congenital heart disease and twinning. Clin Dysmorphol. 1995 Apr;4(2):150-5. PMID 7606322
- [Background] Correa-Villasenor A, Ferencz C, Neill CA, Wilson PD, Boughman JA. Ebstein's malformation of the tricuspid valve: genetic and environmental factors. The Baltimore-Washington Infant Study Group. Teratology. 1994 Aug;50(2):137-47. doi: 10.1002/tera.1420500208. PMID 7801301
- [Background] Ferencz C, Boughman JA. Congenital heart disease in adolescents and adults. Teratology, genetics, and recurrence risks. Cardiol Clin. 1993 Nov;11(4):557-67. PMID 8252559
- [Background] Wilson PD, Correa-Villasenor A, Loffredo CA, Ferencz C. Temporal trends in prevalence of cardiovascular malformations in Maryland and the District of Columbia, 1981-1988. The Baltimore-Washington Infant Study Group. Epidemiology. 1993 May;4(3):259-65. PMID 8512990
- [Background] Rubin JD, Ferencz C, Loffredo C. Use of prescription and non-prescription drugs in pregnancy. The Baltimore-Washington Infant Study Group. J Clin Epidemiol. 1993 Jun;46(6):581-9. doi: 10.1016/0895-4356(93)90132-k. PMID 8501486
- [Background] Kuehl KS, Loffredo CA, Ferencz C. Failure to diagnose congenital heart disease in infancy. Pediatrics. 1999 Apr;103(4 Pt 1):743-7. doi: 10.1542/peds.103.4.743. PMID 10103296
- [Background] Correa-Villasenor A, Ferencz C, Loffredo C, Magee C. Paternal exposures and cardiovascular malformations. The Baltimore-Washington Infant Study Group. J Expo Anal Environ Epidemiol. 1993;3 Suppl 1:173-85. PMID 9857303
- [Background] Wilson PD, Loffredo CA, Correa-Villasenor A, Ferencz C. Attributable fraction for cardiac malformations. Am J Epidemiol. 1998 Sep 1;148(5):414-23. doi: 10.1093/oxfordjournals.aje.a009666. PMID 9737553
- [Background] Rosenthal GL. Patterns of prenatal growth among infants with cardiovascular malformations: possible fetal hemodynamic effects. Am J Epidemiol. 1996 Mar 1;143(5):505-13. doi: 10.1093/oxfordjournals.aje.a008771. PMID 8610666
- [Background] Loffredo CA, Silbergeld EK, Ferencz C, Zhang J. Association of transposition of the great arteries in infants with maternal exposures to herbicides and rodenticides. Am J Epidemiol. 2001 Mar 15;153(6):529-36. doi: 10.1093/aje/153.6.529. PMID 11257060